CLINICAL TRIAL: NCT01376908
Title: A Phase IIIb, Multicentre, Open-Label, Randomized, Controlled Study of the Efficacy, Safety, and Population Pharmacokinetics of Sapropterin Dihydrochloride (Kuvan®) in Phenylketonuria (PKU) Patients <4 Years Old.
Brief Title: Kuvan® in Phenylketonuria Patients Less Than 4 Years Old
Acronym: SPARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700773-003; 2009-015768-33 (EudraCT Number)
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria (PKU); Kuvan® (Sapropterin); Phe-restricted diet; Paediatric <4 years old; responders to BH4; Phe tolerance
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin; Phenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kuvan® + Phe-restricted diet (Experimental): Subjects will be treated with Kuvan® tablets once daily along with Phe-restricted diet therapy.
  Interventions: Drug: Kuvan®; Other: Phenylalanine (Phe)-restricted diet
- Phe-restricted diet alone (Other): Subjects will follow a Phe-restricted diet alone.
  Interventions: Other: Phenylalanine (Phe)-restricted diet

INTERVENTIONS:
Drug: Kuvan® — Kuvan® (sapropterin dihydrochloride) tablets will be administered orally at the dose of 10 mg/kg/day and will be escalated to 20 mg/kg/day if after 4 weeks a subject's Phe tolerance is not increased by at least 20% versus baseline.
  Other Names: Sapropterin dihydrochloride
  Arms: Kuvan® + Phe-restricted diet
Other: Phenylalanine (Phe)-restricted diet — Phe intake will be adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.

SUMMARY:
This is a Phase 3b, multicenter, open-label, randomized, controlled study to evaluate efficacy, safety and population pharmacokinetics of sapropterin dihydrochloride (Kuvan®) in less than 4 year-old infants and children with phenylketonuria (PKU).

ELIGIBILITY:
Inclusion Criteria:

* Male or female PKU infants and young children less than (<) 4 years of age at the scheduled Day 1 visit of the 26-week study period (taking into consideration the maximum of 21 days in the screening period)
* Confirmed clinical and biochemical PKU, including at least two previous blood Phe levels greater than or equal to (>=) 400 micromol per liter (mcmol/L) obtained on 2 separate occasions
* Previously responded, as assessed by the Investigator, to a tetrahydrobiopterin (BH4) test, if all 3 of the following criteria are satisfied:

  1. The BH4 dose was 20 milligram per kilogram per day (mg/kg/day)
  2. The duration of the test was at least for 24 hours
  3. A 30% decrease in blood Phe levels.
* Defined level of dietary Phe tolerance consistent with the diagnosis of PKU
* Good adherence to dietary treatment, including prescribed dietary Phe restriction and prescribed amounts of Phe-free protein supplements and low-Phe foods
* Maintenance of blood Phe levels within the therapeutic target range of 120-360 mcmol/L (defined as >=120 to <360 mcmol/L) over a 4-month period prior to Screening, as assessed by the Investigator
* Parent(s) and/or guardian(s) willing to comply with all study procedures, maintain strict adherence to the diet, and willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any study procedures

Exclusion Criteria:

* Use of Kuvan®, Biopten®, or any unregistered preparation of tetrahydrobiopterin within the previous 30 days, unless for the purposes of a BH4 responsiveness test
* Previous exposure to Kuvan®, Biopten®, or any unregistered preparation of tetrahydrobiopterin for greater than (>)30 days
* Known hypersensitivity to Kuvan® or its excipients
* Known hypersensitivity to other approved or non-approved formulations of tetrahydrobiopterin
* Previous diagnosis of BH4 deficiency
* Current use of methotrexate, trimethoprim, or other dihydrofolate reductase inhibitors
* Current use of medications that are known to affect nitric oxide synthesis, metabolism or action
* Current use of levodopa
* Current use of experimental/other investigational or unregistered drugs that may affect the study outcomes
* Inability to comply with study procedures
* Inability to tolerate oral intake
* History of organ transplantation
* Concurrent disease or condition that would interfere with study participation or increase the risk for adverse events, including seizure disorders, corticosteroid administration, active malignancy, diabetes mellitus, severe congenital heart disease, renal or hepatic failure
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial
* Any condition that, in the view of the Principal Investigator renders the subject at high risk for failure to comply with treatment or to complete the study

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2014-07 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Alvarez, MD, Study Director — BioMarin Pharmaceutical
Locations (22):
- Austria (2):
  - Research Site, Graz
  - Research site, Innsbruck
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Edegem
- Research Site, Prague, Czechia
- Germany (4):
  - Research site, Heidelberg
  - Research Site, Munich
  - Research Site, Münster
  - Research Site, Reutlingen
- Italy (5):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
  - Research site, Rome
- Netherlands (2):
  - Research Site, Amsterdam
  - Research Site, Maastricht
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
- Research Site, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Research Site, Birmingham
  - Research site, London

REFERENCES:
- [Derived] Muntau AC, Burlina A, Eyskens F, Freisinger P, Leuzzi V, Sivri HS, Gramer G, Pazdirkova R, Cleary M, Lotz-Havla AS, Lane P, Alvarez I, Rutsch F. Long-term efficacy and safety of sapropterin in patients who initiated sapropterin at < 4 years of age with phenylketonuria: results of the 3-year extension of the SPARK open-label, multicentre, randomised phase IIIb trial. Orphanet J Rare Dis. 2021 Aug 3;16(1):341. doi: 10.1186/s13023-021-01968-1. PMID 34344399
- [Derived] Muntau AC, Burlina A, Eyskens F, Freisinger P, De Laet C, Leuzzi V, Rutsch F, Sivri HS, Vijay S, Bal MO, Gramer G, Pazdirkova R, Cleary M, Lotz-Havla AS, Munafo A, Mould DR, Moreau-Stucker F, Rogoff D. Efficacy, safety and population pharmacokinetics of sapropterin in PKU patients <4 years: results from the SPARK open-label, multicentre, randomized phase IIIb trial. Orphanet J Rare Dis. 2017 Mar 9;12(1):47. doi: 10.1186/s13023-017-0600-x. PMID 28274234

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 109 subjects screened for the study, 77 pharmacogenetics (PGx) informed consent forms were signed and 73 samples were analyzed which were used as analysis population for outcome measure 11 "Number of samples with phenylalanine hydroxylase (PAH) gene mutations".
Groups:
- Kuvan® + Phe-restricted Diet: Kuvan® (sapropterin dihydrochloride) tablets were administered orally at a dose of 10 milligram/kilogram/day (mg/kg/day). If after 4 weeks, there was less than 20 percent (%) increase in subject's Phe tolerance versus baseline, the dose was escalated to 20 mg/kg/day. Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.
- Phe-restricted Diet: Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.
Period: Overall Study
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Started | 27 | 29
Completed | 25 | 26
Not Completed | 2 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population consisted of all the randomized subjects at the start of the study and were analyzed according to the group allocated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: months] | 21.1 (12.3) | 21.2 (12.0) | 21.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Dietary Phenylalanine (Phe) Tolerance at Week 26
Description: Phe tolerance was defined as the amount of dietary Phe prescribed (milligram per kilogram per day [mg/kg/day]) while maintaining blood Phe levels within the selected therapeutic target range (defined as greater than or equal to [>=] 120 to less than [<] 360 micromoles per liter [mcmol/L]).
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: mg/kg/day
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
mg/kg/day | 80.6 (4.2) | 50.1 (4.3)

2. Secondary Outcome: Mean Blood Phe Levels
Description: Mean blood phe levels were defined as the mean of blood phe levels assessed over each 2-week intervals
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, and 26
Population: Intention-to-treat (ITT) population consisted of all the randomized subjects at the start of the study and were analyzed according to the group allocated. 'n' signifies number of subjects evaluable for this measure at given time points for each reporting group respectively.
Measure: Mean (Standard Deviation); unit: micromol per liter (mmol/L)
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
micromol per liter (mmol/L)
  Baseline (n=27, 29) | 287.3 (166.6) | 352.9 (219.9)
  Week 2 (n=27, 26) | 214.3 (89.3) | 321.3 (133.5)
  Week 4 (n=27, 24) | 202.1 (79.3) | 308.0 (122.2)
  Week 6 (n=25, 26) | 248.0 (85.4) | 303.8 (87.4)
  Week 8 (n=26, 26) | 268.7 (107.9) | 318.0 (108.9)
  Week 10 (n=24, 27) | 271.1 (109.4) | 325.4 (106.2)
  Week 12 (n=22, 22) | 317.6 (106.0) | 328.9 (125.0)
  Week 14 (n=24, 26) | 271.6 (79.0) | 311.2 (118.6)
  Week 16 (n=25, 26) | 320.3 (112.2) | 356.3 (99.1)
  Week 18 (n=24, 26) | 302.9 (122.7) | 325.4 (80.4)
  Week 20 (n=25, 25) | 305.1 (116.1) | 326.3 (77.0)
  Week 22 (n=25, 24) | 293.2 (86.8) | 346.9 (97.8)
  Week 24 (n=24, 25) | 278.8 (77.2) | 326.1 (120.4)
  Week 26 (n=21, 22) | 300.1 (115.2) | 343.3 (118.4)

3. Secondary Outcome: Change From Baseline in Dietary Phe Tolerance After 26 Weeks
Description: Phe tolerance was defined as the amount of dietary Phe ingested (mg/kg/day) while maintaining blood Phe levels within the selected therapeutic target range (defined as >=120 to <360 mcmol/L).
Time Frame: Baseline and at Week 26 (last observation carried-forward [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mg/kg/day
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
mg/kg/day
  Baseline (n=27, 29) | 37.1 (17.3) | 35.8 (20.9)
  Week 26:LOCF (n=27, 27) | 74.0 (38.6) | 49.8 (24.2)
  Change at Week 26: LOCF (n=27, 27) | 36.9 (27.3) | 13.1 (19.6)

4. Secondary Outcome: Number of Subjects With Any TEAEs, AEs Related to Kuvan, Serious AEs, AEs Leading to Death, and AEs Leading to Discontinuation
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study treatment and up to 31 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study drug administration up to 31 days after the last dose of study drug administration
Population: Safety population included all subjects who either received at least one dose of Kuvan in the study period, or were randomized to Phe-restricted diet alone and who had some safety assessment data available.
Measure: Number; unit: subjects
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 27
subjects
  TEAEs | 27 | 27
  AEs related to Kuvan | 8 | 0
  SAEs | 3 | 1
  AEs leading to death | 0 | 0
  AEs Leading to discontinuation | 0 | 0

5. Secondary Outcome: Number of Subjects With Normal Neuromotor Developmental Milestones Assessed Using Denver Developmental Scale (DDS)
Description: Subjects with normal neuromotor development were assessed by standardized developmental milestones using a parent/guardian report form in the following areas: fine motor, gross motor, language, and personal-social using DDS Test. DDS Test is a widely used to examine the developmental progress of 0-6 years of children. The scale reflects what percentage of a certain age group is able to perform a certain task. Tasks are grouped into 4 categories (social contact, fine motor skill, language, and gross motor skill) and include items such as smiles spontaneously (performed by 90% of three-month-olds), knocks 2 building blocks against each other (90% of 13-month-olds), speaks 3 words other than "mom" and "dad" (90% of 21-month-olds), or hops on 1 leg (90% of 5-year-olds). The more items a child fails to perform (passed by 90% of his/her peers), the more likely the child manifests a significant developmental problems.
Time Frame: Baseline, Weeks 12, 26
Population: Intention-to-Treat (ITT) population consisted of all subjects who were randomized at the start of the Study Period and analyzed according to the group allocated. "n" signifies number of evaluable subjects in the specified categories, for each reporting group, respectively.
Measure: Number; unit: subjects
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
subjects
  Fine motor: Baseline (n=25, 26) | 18 | 21
  Fine motor: Week 12 (n=25, 25) | 21 | 23
  Fine motor: Week 26 (n=25, 25) | 20 | 23
  Gross motor: Baseline (n=25, 26) | 23 | 23
  Gross motor: Week 12 (n=25, 25) | 21 | 20
  Gross motor: Week 26 (n=25, 25) | 20 | 19
  Language: Baseline (n=25, 26) | 22 | 20
  Language: Week 12 (n=25, 25) | 22 | 22
  Language: Week 26 (n=25, 25) | 16 | 20
  Personal social: Baseline (n= 25, 26) | 22 | 22
  Personal social: Week 12 (n=25, 25) | 22 | 21
  Personal social: Week 26 (n=25, 25) | 22 | 18

6. Secondary Outcome: Neurodevelopmental Status Assessed Using Bayley III Scales of Infant and Toddler Development
Description: Neurodevelopmental assessments was done using the following age-dependent scales: Bayley III for subjects less than (<) 3.5 years of age and WPPSI III for subjects greater than or equal to (>=) 3.5 to <4 years of age, based on following scores: adaptive behavior composite (ABC) score, cognitive composite (CC) score, language composite (LC) score, motor composite (MC) score., and social-emotional composite (SEC) score. Composite scores ranged from 40 (very poor) to 160 (excellent) and are classified as following: >=115: accelerated performance; 85-114: development within normal limits; 70-84: mildly delayed development; less than or equal to (<=) 69: significant delayed development.
Time Frame: Baseline and Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
Units on a scale
  ABC score: Baseline (n=15, 18) | 106.5 (14.2) | 96.2 (14.6)
  ABC score: Week 26 (n=19, 18) | 102.4 (16.4) | 93.4 (14.1)
  CC score: Baseline (n=19, 20) | 100.0 (11.8) | 101.2 (15.9)
  CC score: Week 26 (n=20, 19) | 102.8 (12.9) | 100.8 (13.0)
  LS score: Baseline (n=18, 19) | 96.7 (12.4) | 97.7 (19.5)
  LS score: Week 26 (n=20, 19) | 98.3 (11.9) | 93.6 (12.1)
  MC score: Baseline (n=19, 20) | 97.8 (13.7) | 94.9 (13.6)
  MC score: Week 26 (n=20, 19) | 100.6 (15.2) | 98.7 (9.5)
  SEC score: Baseline (n=17, 18) | 102.9 (11.3) | 106.0 (16.3)
  SEC score: Week 26 (n=19, 18) | 106.3 (19.1) | 102.5 (13.2)

7. Secondary Outcome: Growth Parameters Standard Deviation Scores (SDS)
Description: Growth assessment was performed by monitoring body mass index, height (or length), weight, and maximal occipital-frontal head circumference (MOFHC). Supine length was measured up to 2 years of age thereafter standing height was measured unless subject was unable to stand upright, in which case supine length was measured. Respective parameter SDS was calculated as the value of parameter minus reference mean value of parameter divided by standard deviation of the reference population.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 26
Population: Intention-to-Treat (ITT) population consisted of all subjects who were randomized at the start of the Study Period and analyzed according to the group allocated. "n" signifies number of evaluable subjects in the specified categories for each reporting group, respectively.
Measure: Mean (Standard Deviation); unit: SDS
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
SDS
  Body mass index SDS: Baseline (n=27, 29) | 0.37 (0.84) | 0.34 (0.99)
  Body mass index SDS: Week 4 (n=26, 27) | 0.33 (0.92) | 0.36 (0.95)
  Body mass index SDS: Week 8 (n=25, 26) | 0.47 (0.93) | 0.38 (0.82)
  Body mass index SDS: Week 12 (n=25, 26) | 0.37 (1.02) | 0.48 (0.91)
  Body mass index SDS: Week 16 (n=25, 26) | 0.34 (0.95) | 0.39 (0.93)
  Body mass index SDS: Week 20 (n=25, 27) | 0.46 (0.93) | 0.44 (0.86)
  Body mass index SDS: Week 26 (n=25, 26) | 0.58 (0.83) | 0.41 (0.81)
  Height SDS: Baseline (n=27, 29) | -0.19 (1.17) | -0.21 (1.03)
  Height SDS: Week 4 (n=26, 27) | -0.19 (1.08) | -0.25 (1.00)
  Height SDS: Week 8 (n=25, 26) | -0.22 (1.08) | -0.13 (1.05)
  Height SDS: Week 12 (n=25, 26) | 0.02 (1.62) | -0.14 (1.11)
  Height SDS: Week 16 (n=25, 26) | 0.05 (1.36) | -0.05 (1.05)
  Height SDS: Week 20 (n=25, 27) | -0.08 (1.21) | -0.11 (0.95)
  Height SDS: Week 26 (n=25, 26) | -0.11 (1.16) | -0.06 (0.92)
  MOFHC SDS: Baseline (n=27, 29) | 0.37 (1.38) | 0.07 (1.10)
  MOFHC SDS: Week 4 (n=25, 26) | 0.48 (1.41) | 0.21 (1.03)
  MOFHC SDS: Week 8 (n=25, 26) | 0.51 (1.40) | 0.35 (1.05)
  MOFHC SDS: Week 12 (n=25, 26) | 0.43 (1.23) | 0.20 (1.19)
  MOFHC SDS: Week 16 (n=25, 26) | 0.58 (1.26) | 0.25 (1.18)
  MOFHC SDS: Week 20 (n=25, 26) | 0.41 (1.30) | 0.18 (1.24)
  MOFHC SDS: Week 26 (n=25, 26) | 0.43 (1.34) | 0.15 (1.26)
  Weight SDS: Baseline (n=27, 29) | 0.12 (0.81) | 0.12 (0.66)
  Weight SDS: Week 4 (n=26, 27) | 0.11 (0.86) | 0.12 (0.64)
  Weight SDS: Week 8 (n=25, 27) | 0.18 (0.88) | 0.18 (0.66)
  Weight SDS: Week 12 (n=25, 26) | 0.23 (0.91) | 0.25 (0.65)
  Weight SDS: Week 16 (n=25, 26) | 0.23 (0.97) | 0.25 (0.74)
  Weight SDS: Week 20 (n=25, 27) | 0.25 (0.95) | 0.24 (0.67)
  Weight SDS: Week 26 (n=25, 26) | 0.32 (0.93) | 0.19 (0.67)

8. Secondary Outcome: Number of Subjects With Hypophenylalanemia
Description: Hypophenylalanemia is defined as the condition of blood Phe levels <120 mcmol/L.
Time Frame: Week 26
Population: Safety population consisted of all subjects who had some safety assessment data available (at least one visit in vital signs, AE or laboratory results) in the Study Period and who received at least one dose of Kuvan in the Study Period, or who were randomized to Phe-restricted diet alone.
Measure: Number; unit: Subjects
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 27
Subjects | 10 | 9

9. Secondary Outcome: Dietary Phe Tolerance During Extension Period
Description: as for outcome 3
Time Frame: Every 6 months during 3 year extension period or until product is commercially approved
Population: The extension period of this study is ongoing. Data will be provided after completion of extension period i.e first quarter 2017
Groups:
- Kuvan® + Phe-restricted Diet: Kuvan® (sapropterin dihydrochloride) tablets were administered orally at a dose of 10 milligram/kilogram/day (mg/kg/day). If after 4 weeks, there was less than 20 percent (%) increase in subject's Phe tolerance versus baseline, the dose was escalated to 20 mg/kg/day. Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.After 26 weeks, the dose may be adjusted by the Investigator, if clinically indicated, but it may not exceed 20 mg/kg/day.
- Phe-restricted Diet: Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria. After 26 weeks, the starting dose of Kuvan will be 10 mg/kg/day, and the dose may be adjusted by the Investigator, if clinically indicated, but it may not exceed 20 mg/kg/day.
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 26
Population: Intention-to-treat (ITT) population consisted of all the randomized subjects at the start of the study and were analyzed according to the group allocated. "n" signifies number of evaluable subjects in the specified categories for each reporting group, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Number analyzed (Participants) | 27 | 29
mmHg
  SBP: Baseline (n=25, 25) | 93.5 (11.0) | 93.1 (14.4)
  SBP: Week 4 (n=22, 25) | 95.9 (14.6) | 101.5 (17.6)
  SBP: Week 8 (n=23, 25) | 95.9 (17.5) | 95.7 (17.9)
  SBP: Week 12 (n=23, 26) | 97.0 (13.2) | 95.2 (9.8)
  SBP: Week 16 (n=23, 26) | 95.0 (14.5) | 98.2 (12.3)
  SBP: Week 20 (n=21, 27) | 95.6 (14.1) | 98.4 (12.6)
  SBP: Week 26 (n=22, 25) | 97.5 (11.1) | 96.8 (8.7)
  DBP: Baseline (n=25, 25) | 55.8 (9.0) | 57.1 (8.1)
  DBP: Week 4 (n=22, 25) | 59.8 (9.8) | 59.0 (13.3)
  DBP: Week 8 (n=23, 25) | 59.1 (7.8) | 55.2 (8.7)
  DBP: Week 12 (n=23, 26) | 58.5 (6.2) | 57.4 (9.7)
  DBP: Week 16 (n=23, 26) | 57.7 (12.1) | 58.5 (11.2)
  DBP: Week 20 (n=21, 27) | 57.5 (12.1) | 58.4 (6.3)
  DBP: Week 26 (n=22, 25) | 59.0 (7.0) | 59.2 (9.4)

11. Secondary Outcome: Number of Samples With Phenylalanine Hydroxylase (PAH) Gene Mutations
Description: The DNA samples received were quantified by using a nanophotometer, and were aliquoted to a concentration of 20 nanogram/microliter DNA and aliquots from each sample were distributed to one 96-well plate. All samples were Sanger sequenced regarding exons 1 to 13 of the PAH gene in forward direction using the DNAs in the 96-well plate. All samples showing variants were Sanger sequenced regarding the concerned exon in reverse direction using DNA from the original tube. All samples showing a homozygous mutation were analyzed by MLPA. All samples showing only 1 mutation were analyzed by MLPA. All samples showing only 1 or no mutation were resequenced completely (exons 1 to 13) in both directions.
Time Frame: Screening (within 42 days prior to Day 1 of the 26-week study period)
Population: Analysis population included subjects who signed pharmacogenetics (PGx) informed consent and whose samples were available for analysis. Out of 109 subjects screened for the study, 77 PGx informed consent forms were signed and 73 samples were analyzed.
Measure: Number; unit: Sample
Groups:
- Pharmacogenetic Evaluation: Kuvan® (sapropterin dihydrochloride) tablets were administered orally at a dose of 10 milligram/kilogram/day (mg/kg/day). If after 4 weeks, there was less than 20 percent (%) increase in subject's Phe tolerance versus baseline, the dose was escalated to 20 mg/kg/day. Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.
Arm/Group | Pharmacogenetic Evaluation
Number analyzed (Participants) | 73
Sample | 73

12. Secondary Outcome: Population Pharmacokinetic (PK) Parameter: Apparent Clearance (CL/f)
Description: CL/f is the rate at which a drug is removed from the body via renal, hepatic and other clearance pathways.The reason for pooling subjects receiving Kuvan and subjects with Phe-restricted Diet was to facilitate the estimation of baseline endogenous value of BH4 which can only be observed in subjects not receiving the treatment. Ignoring this baseline endogenous value would have led to biased stimated of the Kuvan PK parameters. This pooling assumes that the addition of Kuvan does not confound the BH4 measurements in these analyses as a consequence the population PK parameters describing the PK of BH4 are the same for the 2 arms and so cannot be presented in terms of per arm/per treatment group based as per the planned analysis.
Time Frame: Weeks 5 to 12
Population: All enrolled subjects for whom at least one adequately documented BH4 concentration value and dose record were included in the population PK analysis. 'N' (number of subjects analyzed) =subjects evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: liter per hour
Groups:
- Population PK Analysis Set: All enrolled subjects for whom at least one adequately documented BH4 concentration value and dose record were included in the population PK analysis. This includes patients receiving either Kuvan® (sapropterin dihydrochloride) tablets were administered orally at a dose of 10 milligram/kilogram/day (mg/kg/day) in conjunction with a Phe-restricted diet, or diet alone. If after 4 weeks, there was less than 20 percent (%) increase in subject's Phe tolerance versus baseline, the Kuvan® dose was escalated to 20 mg/kg/day. Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 52
liter per hour | 2780 (2)

13. Secondary Outcome: Population PK Parameter: Apparent Volume of Distribution (V/f)
Description: V/f is defined as the distribution of a medication between the plasma and the rest of the body after the dose. It is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of the drug. The reason for pooling subjects receiving Kuvan and subjects with Phe-restricted Diet was to facilitate the estimation of baseline endogenous value of BH4 which can only be observed in subjects not receiving the treatment. Ignoring this baseline endogenous value would have led to biased stimated of the Kuvan PK parameters. This pooling assumes that the addition of Kuvan does not confound the BH4 measurements in these analyses as a consequence the population PK parameters describing the PK of BH4 are the same for the 2 arms and so cannot be presented in terms of per arm/per treatment group based as per the planned analysis.
Time Frame: Weeks 5 to 12
Population: as for outcome 12
Measure: Mean (Standard Error); unit: liter
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 52
liter | 3870 (5.9)

14. Secondary Outcome: Population PK Parameter: Area Under the Plasma Concentration Curve, Time 0 to Infinity (AUC [0-infinity])
Description: AUC [0-infinity] was estimated by determining total area under the curve of the concentration versus time curve extrapolated to infinity. Since AUC could not be obtained from non-compartmental analysis because of sparse data, AUC = Dose/(CL/F); CL/F was population apparent clearance estimated from the population PK model, & Dose the actual total dose received by the patient on one dosing interval. The reason for pooling subjects receiving Kuvan &subjects with Phe-restricted Diet was to facilitate estimation of baseline endogenous value of BH4 which can only be observed in subjects not receiving treatment. Ignoring this baseline endogenous value would have led to biased estimated of Kuvan PK parameters. This pooling assumes that the the addition of Kuvan does not confound the BH4 measurements in these analyses as a consequence the population PK parameters describing the PK of BH4 were same for the 2 arms and cannot be presented per arm/per treatment group as per planned analysis.
Time Frame: Weeks 5 to 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram*hour per liter(mcg*hour/liter)
Groups:
- Population PK Analysis Set: Age Group 1 (< 1 Year); Population PK Analysis Set: Age Group 2 (1 to 2 Years); Population PK Analysis Set: Age Group 2 (>= 2 Years): All enrolled subjects for whom at least one adequately documented BH4 concentration value and dose record were included in the population PK analysis. This includes patients receiving either Kuvan® (sapropterin dihydrochloride) tablets were administered orally at a dose of 10 milligram/kilogram/day (mg/kg/day) in conjunction with a Phe-restricted diet, or diet alone. If after 4 weeks, there was less than 20 percent (%) increase in subject's Phe tolerance versus baseline, the Kuvan® dose was escalated to 20 mg/kg/day. Phenylalanine (Phe)-restricted diet was adjusted every 2 weeks, based on the mean Phe levels of the previous 2 weeks using pre-defined Phe adjustment criteria.
Arm/Group | Population PK Analysis Set: Age Group 1 (< 1 Year) | Population PK Analysis Set: Age Group 2 (1 to 2 Years) | Population PK Analysis Set: Age Group 2 (>= 2 Years)
Number analyzed (Participants) | 14 | 18 | 20
microgram*hour per liter(mcg*hour/liter) | 234.89 (89.82) | 215.74 (63.88) | 206.22 (103.24)

15. Secondary Outcome: Population PK Parameter: Terminal Elimination Half-life (t1/2)
Description: The t1/2 was defined as the time required for plasma concentration of drug to decrease 50 percent (%) in the final stage of elimination. Since t1/2 could not be obtained from non-compartmental analysis because of sparse data, t1/2 was estimated as Log(2)*(V/F)/(CL/F), where V/F & CL/F were the population apparent central Volume & clearance, estimated from population PK model. The reason for pooling subjects receiving Kuvan & subjects with Phe-restricted Diet was to facilitate the estimation of baseline endogenous value of BH4 which can only observed in subjects not receiving treatment. Ignoring this baseline endogenous value would have led biased stimated of the Kuvan PK parameters. This pooling assumes that the addition of Kuvan does not confound the BH4 measurements in these analyses as a consequence the population PK parameters describing the PK of BH4 are the same for the 2 arms and so cannot be presented in terms of per arm/per treatment group based as per the planned analysis.
Time Frame: Weeks 5 to 12
Population: as for outcome 12
Measure: Number; unit: hours
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 52
hours | 0.96

16. Secondary Outcome: Population PK Parameter: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Up to Week 26
Population: Cmax could not be calculated from the model derived parameters because shrinkage was over 20% for V/f and interindividual variability could not be estimated for absorption rate constant (Ka).
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 0

17. Secondary Outcome: Population PK Parameter: Time to Maximum Plasma Concentration (Tmax)
Time Frame: Up to Week 26
Population: Tmax could not be calculated from the model derived parameters because shrinkage was over 20% for V/F and interindividual variability could not be estimated for Ka.
Arm/Group | Population PK Analysis Set
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration up to 31 days after the last dose of study drug administration
Description: Safety population included all subjects who either received at least one dose of Kuvan in the study period, or were randomized to Phe-restricted diet alone and who had some safety assessment data available.
Arm/Group | Kuvan® + Phe-restricted Diet | Phe-restricted Diet
Serious Adverse Events (participants affected / at risk) | 3/27 | 1/27
Other Adverse Events (participants affected / at risk) | 26/27 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan® + Phe-restricted Diet (N=27) | Phe-restricted Diet (N=27)
Gastroenteritis (Infections and infestations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kuvan® + Phe-restricted Diet (N=27) | Phe-restricted Diet (N=27)
Nasopharyngitis (Infections and infestations) | 13 | 11
Rhinitis (Infections and infestations) | 8 | 6
Pharyngitis (Infections and infestations) | 7 | 3
Gastroenteritis (Infections and infestations) | 3 | 3
Otitis media (Infections and infestations) | 2 | 3
Bronchitis (Infections and infestations) | 2 | 2
Pyrexia (General disorders) | 17 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 10 | 9
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Abdominal Pain (Gastrointestinal disorders) | 3 | 2
Amino acid level decreased (Investigations) | 10 | 9
Rash (Skin and subcutaneous tissue disorders) | 5 | 2
Conjunctivitis (Eye disorders) | 2 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other